CLINICAL TRIAL: NCT02761057
Title: A Randomized, Phase II Efficacy Assessment of Multiple MET Kinase Inhibitors (Cabozantinib [NSC #761968], Crizotinib [NSC #749005], Savolitinib [NSC #785348], and Sunitinib [NSC #736511]) in Metastatic Papillary Renal Carcinoma (PAPMET)
Brief Title: Testing Cabozantinib, Crizotinib, Savolitinib and Sunitinib in Kidney Cancer Which Has Progressed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01707; NCI-2015-01707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1500 (Other: SWOG); S1500 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Results first posted 2022-09-02 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Papillary Renal Cell Carcinoma; Metastatic Papillary Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7; Type 1 Papillary Renal Cell Carcinoma; Type 2 Papillary Renal Cell Carcinoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; cabozantinib; Crizotinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (sunitinib malate) (Experimental): Patients receive sunitinib malate PO QD on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Sunitinib Malate
- Arm II (cabozantinib s-malate) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography
- Arm III (crizotinib closed to accrual 12/5/18) (Experimental): Patients receive crizotinib PO BID on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Crizotinib
- Arm IV (savolitinib closed to accrual 12/5/18) (Experimental): Patients receive savolitinib PO QD on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Savolitinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of plasma and serum samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm II (cabozantinib s-malate)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Crizotinib — Given PO
  Other Names: Alkixen; Crizocent; MET Tyrosine Kinase Inhibitor PF-02341066; PF 02341066; PF-02341066; PF-2341066; PF02341066; Xalkori
  Arms: Arm III (crizotinib closed to accrual 12/5/18)
Drug: Savolitinib — Given PO
  Other Names: AZD 6094; AZD6094; HMPL-504; Volitinib
  Arms: Arm IV (savolitinib closed to accrual 12/5/18)
Drug: Sunitinib Malate — Given PO
  Other Names: SU 011248; SU 11248; SU-011248; SU-11248; SU011248; SU11248; sunitinib; Sutent
  Arms: Arm I (sunitinib malate)

SUMMARY:
This phase II trial studies how well cabozantinib s-malate, crizotinib, savolitinib, or sunitinib malate work in treating patients with kidney cancer that has spread from where it started to nearby tissue or lymph nodes or to other places in the body. Cabozantinib s-malate, crizotinib, savolitinib, and sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving cabozantinib s-malate, crizotinib, or savolitinib will work better in treating patients with kidney cancer compared to sunitinib malate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) in patients with metastatic papillary renal cell carcinoma (mPRCC) treated with sunitinib malate (sunitinib) to PFS in patients with mPRCC treated with MET kinase inhibitors.

SECONDARY OBJECTIVES:

I. To compare Response Evaluation Criteria in Solid Tumors (RECIST) response rate (RR; defined as the combined rate of confirmed and unconfirmed partial response [PR] and confirmed and unconfirmed complete response [CR]) in patients with mPRCC treated with sunitinib to RR in patients treated with putative MET inhibitors.

II. To compare overall survival (OS) in patients with mPRCC treated with sunitinib to OS in patients with mPRCC treated with putative MET inhibitors.

III. To compare the safety profile of sunitinib and putative MET inhibitors in patients with mPRCC.

TRANSLATIONAL OBJECTIVES:

I. To evaluate the prognostic and predictive value of MET mutations, MET copy number or other markers of MET signaling in patients with mPRCC treated with putative MET inhibitors.

II. To estimate the frequency of high oncometabolite levels in formalin-fixed, paraffin-embedded (FFPE) tissues of patients with advanced papillary renal cell carcinoma by liquid chromatography-mass spectrometry (LC-MS/MS) and estimate progression free survival for those with and without high oncometabolite levels being treated.

III. To correlate the mutational signature suggestive of a homologous recombination defect with high oncometabolite levels in patients with papillary renal cell carcinoma pRCC.

OUTLINE: Patients are randomized to 1 of 4 treatment arms. As of 12/5/18, patients will only be randomized to Arm I or Arm II.

ARM I: Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.

ARM II: Patients receive cabozantinib s-malate PO QD on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.

ARM III (CLOSED TO ACCRUAL 12/5/18): Patients receive crizotinib PO twice daily (BID) on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.

ARM IV (CLOSED TO ACCRUAL 12/5/18): Patients receive savolitinib PO QD on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT at screening and on study, undergo bone scan as clinically indicated, and undergo collection of plasma and serum samples at screening, on study, and during follow up.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary histology renal cell carcinoma which is metastatic or locally advanced disease not amenable to surgical resection; (NOTE: a designation of type I or type II should be made by the local pathologist if possible); mixed histologies containing type I or type II will be allowed provided that they contain >= 50% of the papillary component
* Patients must also have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension; disease X-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; if there is clinical suspicion for bone metastases at the time of enrollment (at the discretion of the investigator), bone scan should be performed at baseline (within 42 days prior to registration); all disease must be assessed and documented on the Baseline Tumor Assessment form
* Patients with a history of treated brain metastases who are asymptomatic and have not received steroid therapy in the 14 days prior to registration are eligible; anti-seizure medications are allowed provided they are non-enzyme inducing (e.g. topiramate, levetiracetam, gabapentin)
* Patients must not have cavitating pulmonary lesions; patients must not have tumor invading the gastrointestinal (GI) tract or evidence of endotracheal or endobronchial tumor within 28 days prior to registration
* Patients may have received prior surgery; at least 28 days must have elapsed since surgery and patient must have recovered from any adverse effects of surgery
* Patients may have received up to one prior systemic therapy for advanced or metastatic renal cell carcinoma with the exception of another VEGF inhibitor Food and Drug Administration (FDA)-approved for advanced renal cell carcinoma (RCC) (i.e., pazopanib, bevacizumab, sorafenib or axitinib); if a patient develops metastatic disease within six months of discontinuation of adjuvant therapy, this will constitute one prior systemic therapy for advanced or metastatic RCC; if a patient develops metastatic disease and more than six months has elapsed since discontinuation of adjuvant therapy, this will not constitute prior systemic therapy for advanced or metastatic RCC; patients may have also received prior immunotherapy; patients must not have received a MET/hepatocyte growth factor (HGF) inhibitor or sunitinib as prior therapy; at least 14 days must have elapsed since completion of prior systemic therapy; patients must have recovered from all associated toxicities at the time of registration
* Patients may have received prior radiation therapy, but must have measurable disease outside the radiation port; at least 14 days must have elapsed since completion of prior radiation therapy; patients must have recovered from all associated toxicities at the time of registration
* Patients must not be taking, nor plan to take while on protocol treatment, strong CYP3A4 inhibitors (e.g. boceprevir, cobicistat, danoprevir, elvitegravir/RIT, fluvoxamine, indinavir, itraconazole, ketoconazole, lopinavir/RIT, nefazodone, nelfinavir, posaconazole, ritonavir, telaprevir, telithromycin, tipravavir/RIT, or voriconazole); strong CYP3A4 inducers (e.g. avasimibe, phenytoin, rifampin, rifabutin); potent inhibitors of CYP1A2 (e.g. ciprofloxacin); and/or drugs known to be CYP3A4 substrates with a narrow therapeutic range (e.g., diergotamine, ergotamine) within 14 days prior to randomization; moderate inhibitors or inducers of isoenzyme CYP3A4 should be avoided, but if necessary can be used with caution
* Patients must not be receiving or planning to receive any other investigational agents
* Patients must have a complete physical examination and medical history within 28 days prior to registration
* Patients must have a Zubrod performance status of 0 - 1
* White blood cell count (WBC) >= 2,000/mcL (must be obtained within 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,000/mcL (must be obtained within 28 days prior to registration)
* Platelet count >= 75,000/mcL (must be obtained within 28 days prior to registration)
* Serum bilirubin =< 1.5 x institutional upper limits of normal (ULN) (must be obtained within 28 days prior to registration)
* Serum transaminase (serum glutamic oxaloacetic transaminase [SGOT]/aspartate aminotransferase [AST] and serum glutamate pyruvate transaminase [SGPT]/alanine aminotransferase [ALT]) must be =< 2.5 x the institutional ULN unless the liver is involved with the tumor, in which case serum transaminase (SGOT/SGPT) must be =< 5 x the institutional ULN (must be obtained within 28 days prior to registration)
* Serum creatinine must be =< 2 x the institutional ULN OR creatinine clearance (either measured or calculated) must be > 30 mL/min (must be obtained within 28 days prior to registration)
* Patients must not have any clinical evidence of congestive heart failure (CHF) (specifically, New York Heart Association [NYHA] class III [moderate] or class IV [severe]) at the time of registration; baseline echocardiogram within 28 days of registration must demonstrate an ejection fraction (EF) >= 50%; due to the potential cardiac toxicity of the agents utilized in this protocol, patients must have corrected QT (QTc) interval < 500 msec on prestudy electrocardiogram (EKG) and no known history of congenital long QT syndrome; patients must not have experienced unstable angina pectoris, clinically significant cardiac arrhythmias, or stroke (transient ischemic attack [TIA] or other ischemic event) within 3 months prior to registration and not have experienced myocardial infarction or thromboembolic event requiring anticoagulation within 6 months of registration; prestudy EKG must be obtained within 28 days prior to registration
* Baseline urinalysis should show urine protein < 3+ and must be obtained within 28 days prior to registration; if urine protein is 3+ or greater, then urine protein by 24 hour collection must show less than 3 grams of protein
* Patients must not have inadequately controlled hypertension; patients must have documented blood pressures of systolic blood pressure (SBP) < 150 and diastolic blood pressure (DBP) < 90 within 14 days of starting randomization; blood pressure medications (any number) are permitted
* Patients must be able to take oral medications (i.e., swallow pills whole); patients must not have gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures that could in the opinion of the treating investigator affect absorption, or active peptic ulcer disease; patients with intractable nausea or vomiting are not eligible
* Patients must not have had any clinically-significant GI bleeding within 6 months prior to registration and patients must not have a GI disorder which (at the discretion of the investigator) bears a high risk of perforation or fistula; examples of this include (but are not limited to) Crohn's disease or tumor with transmural extension through the gastrointestinal lining
* Patients must not have had hemoptysis of >= 0.5 teaspoon (2.5 ml) of red blood within 3 months prior registration
* Patients must not demonstrate any other signs indicative of pulmonary hemorrhage within 3 months prior to registration
* Patient's baseline imaging must not indicate the presence of tumor invading or encasing any major blood vessels
* Patients must not have any unresolved wounds from previous surgery
* Albumin, alkaline phosphatase, bicarbonate, blood urea (BUN), chloride, glucose, phosphorus, and total protein must be assessed within 28 days of registration
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for 3 years; men receiving active surveillance for prostate cancer may also be enrolled
* Due to the unknown effects of the study drugs, patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method while receiving study drug and for three months after last dose of study drug; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cabozantinib, crizotinib, savolitinib or sunitinib; in addition these patients are at increased risk of lethal infections when treated with marrow suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients must be >= 18 years of age
* Patients must have tissue available and be willing to submit for independent pathologic review in order to classify type I versus type II papillary disease
* Patients must be offered the opportunity to participate in specimen banking for future translational medicine studies
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — SWOG Cancer Research Network
Locations (595):
- United States (586):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Research Alliance, Albuquerque, New Mexico
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Saint Joseph's Healthcare Charlton Campus, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] Barata P, Tangen C, Plets M, Thompson IM Jr, Narayan V, George DJ, Heng DYC, Shuch B, Stein M, Gulati S, Tretiakova M, Tripathi A, Bjarnason GA, Humphrey P, Adeniran A, Vaishampayan U, Alva A, Zhang T, Cole S, Lara PN Jr, Lerner SP, Balzer-Haas N, Pal SK. Final Overall Survival Analysis of S1500: A Randomized, Phase II Study Comparing Sunitinib With Cabozantinib, Crizotinib, and Savolitinib in Advanced Papillary Renal Cell Carcinoma. J Clin Oncol. 2024 Nov 20;42(33):3911-3916. doi: 10.1200/JCO.24.00767. Epub 2024 Sep 10. PMID 39255440
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Pal SK, Tangen C, Thompson IM Jr, Balzer-Haas N, George DJ, Heng DYC, Shuch B, Stein M, Tretiakova M, Humphrey P, Adeniran A, Narayan V, Bjarnason GA, Vaishampayan U, Alva A, Zhang T, Cole S, Plets M, Wright J, Lara PN Jr. A comparison of sunitinib with cabozantinib, crizotinib, and savolitinib for treatment of advanced papillary renal cell carcinoma: a randomised, open-label, phase 2 trial. Lancet. 2021 Feb 20;397(10275):695-703. doi: 10.1016/S0140-6736(21)00152-5. Epub 2021 Feb 13. PMID 33592176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 152 participants were enrolled and randomly assigned. Five participants were excluded because of inadequate baseline disease assessment or no evidence of metastatic disease. Therefore, 147 were deemed eligible and analyzable for the primary analysis.
Groups:
- Arm I (Sunitinib Malate): Patients receive sunitinib malate PO on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Sunitinib Malate: Given PO
- Arm II (Cabozantinib S-malate): Patients receive cabozantinib s-malate PO on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Arm III (Crizotinib Closed to Accrual 12/5/18): Patients receive crizotinib PO BID on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Crizotinib: Given PO
- Arm IV (Savolitinib Closed to Accrual 12/5/18): Patients receive savolitinib PO on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Savolitinib: Given PO
Period: Overall Study
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Cabozantinib S-malate) | Arm III (Crizotinib Closed to Accrual 12/5/18) | Arm IV (Savolitinib Closed to Accrual 12/5/18)
Started | 48 | 46 | 28 | 30
Eligible | 46 | 44 | 28 | 29
Received Protocol Treatment | 45 | 43 | 27 | 28
Completed | 0 | 0 | 0 | 0
Not Completed | 48 | 46 | 28 | 30
Not completed — Ineligible - No Measurable Disease | 1 | 1 | 0 | 1
Not completed — Ineligible - Inadequate Baseline Disease Assessment | 1 | 1 | 0 | 0
Not completed — Currently On Study Treatment | 0 | 3 | 0 | 0
Not completed — Adverse Event | 11 | 9 | 5 | 3
Not completed — Refusal Unrelated to Adverse Event | 2 | 2 | 0 | 2
Not completed — Progression/Relapse | 29 | 27 | 20 | 23
Not completed — Death | 2 | 2 | 1 | 1
Not completed — Other - Not Protocol Specified | 2 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included only eligible participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Cabozantinib S-malate) | Arm III (Crizotinib Closed to Accrual 12/5/18) | Arm IV (Savolitinib Closed to Accrual 12/5/18) | Total
Number analyzed (Participants) | 46 | 44 | 28 | 29 | 147
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [58 to 73] | 65 [58 to 75] | 68 [61 to 75] | 67 [58 to 72] | 66 [58 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 6 | 10 | 35
  Male | 35 | 36 | 22 | 19 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 46 | 40 | 26 | 24 | 136
  Unknown or Not Reported | 0 | 2 | 1 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 9 | 4 | 3 | 21
  White | 39 | 32 | 22 | 21 | 114
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 1 | 3 | 6
Previous Systemic Therapy [Count of Participants; unit: Participants] | 3 | 2 | 2 | 3 | 10
Histological Subtype (Local Assessment) [Count of Participants; unit: Participants] — Papillary renal cell carcinoma (pRCC) histological subtype as determined by a local pathologist. Type 1 is characterized by small cells in a a single layer with scant basophilic cytoplasm and oval nuclei. Type 2 is characterized by large cells with eosinophilic cytoplasm and spherical nuclei with prominent nucleoli and pseudostratification. Type 1 is more common and grows slowly and type 2 is more aggressive and grows more quickly. In general, type 2 pRCC has a poorer prognosis than type 1.
  Participants
    Type 1 | 8 | 9 | 5 | 5 | 27
    Type 2 | 24 | 25 | 15 | 15 | 79
    Not otherwise specified | 14 | 10 | 8 | 9 | 41
Histological Subtype (Central Assessment) [Count of Participants; unit: Participants] — Papillary renal cell carcinoma (pRCC) histological subtype as determined by a central pathologic assessment. Type 1 is characterized by small cells in a a single layer with scant basophilic cytoplasm and oval nuclei. Type 2 is characterized by large cells with eosinophilic cytoplasm and spherical nuclei with prominent nucleoli and pseudostratification. Type 1 is more common and grows slowly and type 2 is more aggressive and grows more quickly. In general, type 2 pRCC has a poorer prognosis than type 1.
  Participants
    Type 1 | 12 | 14 | 9 | 6 | 41
    Type 2 | 21 | 16 | 13 | 13 | 63
    Mixed or Other | 11 | 12 | 5 | 7 | 35
    Missing | 2 | 2 | 1 | 3 | 8
IMDC Risk Group [Count of Participants; unit: Participants] — The International Metastatic Renal Cell Carcinoma Database Consortium's (IMDC) prognostic model to predict survival of metastatic kidney cancer patients has become the standard model used in clinical trials to categorize patients into favorable, intermediate, and poor risk based on treatment time, performance status, and hemoglobin, calcium, neutrophil, and platelet counts.
  Participants
    Favourable | 14 | 10 | 8 | 6 | 38
    Intermediate | 26 | 28 | 16 | 19 | 89
    High | 6 | 6 | 4 | 4 | 20
Zubrod Performance Score [Count of Participants; unit: Participants] — Zubrod performance status scores range from 0 to 4, with higher scores reflecting greater disability. This study only includes participants with a score of 0-1.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 29 | 29 | 18 | 15 | 91
    1 | 17 | 15 | 10 | 14 | 56
Previous Nephrectomy [Count of Participants; unit: Participants] | 34 | 32 | 26 | 21 | 113
Metastatic Sites of Interest [Count of Participants; unit: Participants]
  Bone | 7 | 6 | 5 | 8 | 26
  CNS | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of appropriate diameters of target lesions over smallest sum observed, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause; assessed up to 3 years
Population: Analysis population included eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sunitinib: Experimental: Arm I (sunitinib malate) Patients receive sunitinib malate PO on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity
  Drug: Sunitinib Malate Given PO
  Other Names:
  SU011248 SU11248 sunitinib Sunitinib Malate Sutent
- Cabozantinib: Experimental: Arm II (cabozantinib s-malate) Patients receive cabozantinib s-malate PO on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Drug: Cabozantinib S-malate Given PO
  Other Names:
  BMS-907351 Cabometyx CABOZANTINIB S-MALATE Cometriq XL-184 XL184
- Crizotinib: Experimental: Arm III (crizotinib closed to accrual 12/5/18) Patients receive crizotinib PO BID on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Drug: Crizotinib Given PO
  Other Names:
  CRIZOTINIB MET Tyrosine Kinase Inhibitor PF-02341066XXPF-02341066 PF-2341066 Xalkori
- Savolitinib: Experimental: Arm IV (savolitinib closed to accrual 12/5/18) Patients receive savolitinib PO on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Drug: Savolitinib Given PO
  Other Names:
  AZD 6094 AZD6094 HMPL-504 SAVOLITINIB Volitinib
Arm/Group | Sunitinib | Cabozantinib | Crizotinib | Savolitinib
Number analyzed (Participants) | 46 | 44 | 28 | 29
months | 5.6 [2.9 to 6.7] | 9.0 [5.6 to 12.4] | 2.8 [2.6 to 3.6] | 3.0 [2.8 to 7.2]
Statistical Analysis 1: Comparison: Sunitinib vs Cabozantinib; A proportional hazards model was used to compare the Hazard Ratio (HR) for PFS; Test type: Superiority; p = 0.019, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.37 to 0.97]

2. Secondary Outcome: Response Rate (RR)
Description: The response rate (RR) is defined as the combined rate of confirmed and unconfirmed partial response and confirmed and unconfirmed complete response. Complete response (CR) is defined as the complete disappearance of all target and non-target lesions, along with no new lesions. Partial response (PR) is defined as >=30% decrease of the sum of appropriate diameters of all target measurable lesions, along with no new lesions.
Time Frame: Up to 3 years
Population: Analysis population included eligible participants.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Cabozantinib | Crizotinib | Savolitinib
Number analyzed (Participants) | 46 | 44 | 28 | 29
percentage of participants | 4.35 | 22.73 | 0 | 3.45
Statistical Analysis 1: Comparison: Sunitinib vs Cabozantinib; The Chi-Square test will be used to compare RR between sunitinib and cabozantinib; Test type: Superiority; p = 0.10, Chi-squared

3. Secondary Outcome: Overall Survival (OS)
Description: Duration from date of randomization to date of death from any cause.
Time Frame: Up to 3 years
Population: Analysis population included eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Cabozantinib | Crizotinib | Savolitinib
Number analyzed (Participants) | 46 | 44 | 28 | 29
months | 16.4 [12.8 to 21.6] | 20.0 [11.3 to NA] — There was not enough data to estimate the upper bound 95% CI | 19.9 [11.2 to NA] — There was not enough data to estimate the upper bound 95% CI | 11.7 [6.7 to 28.9]
Statistical Analysis 1: Comparison: Sunitinib vs Cabozantinib; The log-rank test will be used to compare OS; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.47 to 1.51]

4. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Eligible participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Sunitinib | Cabozantinib | Crizotinib | Savolitinib
Number analyzed (Participants) | 45 | 43 | 27 | 28
Participants
  Abdominal pain | 1 | 3 | 0 | 0
  Acute kidney injury | 1 | 0 | 0 | 0
  Alanine aminotransferase increased | 1 | 1 | 2 | 0
  Allergic reaction | 0 | 0 | 1 | 0
  Anemia | 6 | 0 | 1 | 0
  Anorexia | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 1 | 0 | 1 | 0
  Back pain | 0 | 1 | 0 | 0
  Confusion | 0 | 1 | 0 | 0
  Dehydration | 1 | 0 | 0 | 1
  Diarrhea | 3 | 2 | 0 | 0
  Duodenal ulcer | 1 | 0 | 0 | 0
  Dyspnea | 0 | 0 | 0 | 1
  Edema limbs | 0 | 0 | 1 | 2
  Epistaxis | 1 | 0 | 0 | 0
  Facial pain | 1 | 0 | 0 | 0
  Fall | 0 | 2 | 0 | 0
  Fatigue | 3 | 6 | 2 | 0
  Febrile neutropenia | 0 | 1 | 0 | 0
  Gastrointestinal disorders - Other, specify | 0 | 1 | 0 | 0
  Generalized muscle weakness | 1 | 0 | 0 | 1
  Genital edema | 0 | 0 | 0 | 1
  Hearing impaired | 0 | 0 | 0 | 1
  Hematoma | 0 | 1 | 0 | 1
  Hypercalcemia | 0 | 1 | 0 | 0
  Hyperkalemia | 0 | 0 | 1 | 0
  Hypermagnesemia | 0 | 1 | 0 | 0
  Hypertension | 9 | 14 | 0 | 1
  Hypoalbuminemia | 1 | 0 | 1 | 0
  Hypocalcemia | 0 | 1 | 0 | 0
  Hypomagnesemia | 0 | 2 | 0 | 0
  Hyponatremia | 2 | 3 | 0 | 3
  Hypophosphatemia | 0 | 6 | 0 | 0
  Hypoxia | 0 | 1 | 0 | 0
  Infections and infestations - Other, specify | 0 | 1 | 0 | 0
  Lung infection | 0 | 1 | 0 | 0
  Lymphedema | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 2 | 0 | 0 | 0
  Lymphocyte count increased | 1 | 0 | 0 | 0
  Mucositis oral | 0 | 1 | 0 | 0
  Muscle weakness lower limb | 0 | 1 | 0 | 0
  Nausea | 4 | 0 | 0 | 0
  Nervous system disorders - Other, specify | 0 | 1 | 0 | 0
  Neutrophil count decreased | 4 | 0 | 0 | 0
  Pain | 1 | 0 | 0 | 0
  Pain in extremity | 0 | 1 | 1 | 0
  Palmar-plantar erythrodysesthesia syndrome | 0 | 9 | 0 | 0
  Pancreatitis | 0 | 1 | 0 | 0
  Paronychia | 0 | 1 | 0 | 0
  Platelet count decreased | 2 | 0 | 0 | 0
  Pleural effusion | 1 | 0 | 0 | 0
  Pneumonitis | 0 | 1 | 0 | 0
  Proteinuria | 1 | 1 | 0 | 0
  Rash maculo-papular | 0 | 0 | 1 | 1
  Renal calculi | 1 | 0 | 0 | 0
  Reproductive system and breast disorders - Other | 0 | 1 | 0 | 0
  Sinus bradycardia | 0 | 0 | 1 | 0
  Sinus tachycardia | 0 | 0 | 1 | 0
  Skin ulceration | 0 | 1 | 0 | 0
  Somnolence | 1 | 0 | 0 | 0
  Syncope | 0 | 0 | 1 | 0
  Thromboembolic event | 0 | 6 | 0 | 2
  Thrombotic thrombocytopenic purpura | 1 | 0 | 0 | 0
  Vascular disorders - Other, specify | 0 | 0 | 0 | 1
  Vomiting | 1 | 0 | 0 | 0
  White blood cell decreased | 5 | 0 | 0 | 0

5. Other Pre Specified Outcome: MET Mutation Rate
Description: The hazard ratio between the MET inhibitor versus (vs.) sunitinib in those with versus without the mutation (i.e., the interaction) will be compared. Response Evaluation Criteria in Solid Tumors (RECIST) response rate (confirmed and unconfirmed partial response and complete response) based on MET mutation/expression level will be compared using the chi-square test.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: 143 participants who received protocol treatment were evaluable for AEs: 45 on sunitinib arm, 43 on cabozantinib arm, 27 on crizotinib arm, and 28 on savolitinib arm. Adverse Events (AEs) are reported by CTCAE Version 4.0 and Serious Adverse Events (SAEs) are reported by CTCAE Version 5.0. All started participants were monitored/assessed for All-Cause Mortality".
Groups:
- Sunitinib: Experimental: Arm I (sunitinib malate) Patients receive sunitinib malate PO on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Drug: Sunitinib Malate Given PO
  Other Names:
  SU011248 SU11248 sunitinib Sunitinib Malate Sutent
- Crizotinib: Experimental: Arm III (crizotinib closed to accrual 12/5/18) Patients receive crizotinib PO BID on days 1-42. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Drug: Crizotinib Given PO
  Other Names:
  CRIZOTINIB MET Tyrosine Kinase Inhibitor PF-02341066 PF-02341066 PF-2341066 Xalkori
Arm/Group | Sunitinib | Cabozantinib | Crizotinib | Savolitinib
All-Cause Mortality (participants affected / at risk) | 24/46 | 22/44 | 16/28 | 21/29
Serious Adverse Events (participants affected / at risk) | 15/45 | 19/43 | 8/27 | 11/28
Other Adverse Events (participants affected / at risk) | 44/45 | 41/43 | 26/27 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=45) | Cabozantinib (N=43) | Crizotinib (N=27) | Savolitinib (N=28)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 1
Fever (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 1 | 0 | 0
Sudden death NOS (General disorders) | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Nervous system disorders-Other (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 5 | 0 | 1
Vascular disorders-Other (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=45) | Cabozantinib (N=43) | Crizotinib (N=27) | Savolitinib (N=28)
Anemia (Blood and lymphatic system disorders) | 17 | 12 | 7 | 7
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 | 5 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 3 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 1 | 0 | 2
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 0 | 1 | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 3 | 6 | 0 | 0
Hypothyroidism (Endocrine disorders) | 8 | 17 | 0 | 0
Blurred vision (Eye disorders) | 2 | 3 | 1 | 0
Eye disorders-Other (Eye disorders) | 0 | 3 | 6 | 0
Flashing lights (Eye disorders) | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 8 | 3 | 7
Bloating (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 13 | 15 | 8 | 4
Diarrhea (Gastrointestinal disorders) | 22 | 25 | 11 | 6
Dry mouth (Gastrointestinal disorders) | 5 | 8 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 2 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 1 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 3 | 7 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 13 | 16 | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 18 | 8 | 15
Vomiting (Gastrointestinal disorders) | 10 | 10 | 3 | 6
Chills (General disorders) | 3 | 1 | 0 | 3
Edema limbs (General disorders) | 7 | 6 | 9 | 12
Fatigue (General disorders) | 30 | 31 | 16 | 16
Fever (General disorders) | 2 | 5 | 2 | 2
General disorders and admin site conditions - Other (General disorders) | 2 | 3 | 1 | 1
Non-cardiac chest pain (General disorders) | 6 | 3 | 1 | 1
Pain (General disorders) | 5 | 8 | 4 | 3
Lung infection (Infections and infestations) | 2 | 4 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 3 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 7 | 14 | 8 | 4
Alkaline phosphatase increased (Investigations) | 6 | 6 | 4 | 10
Aspartate aminotransferase increased (Investigations) | 9 | 17 | 7 | 4
Blood bilirubin increased (Investigations) | 3 | 2 | 0 | 3
Creatinine increased (Investigations) | 16 | 8 | 10 | 10
Investigations-Other (Investigations) | 4 | 6 | 1 | 1
Lymphocyte count decreased (Investigations) | 12 | 6 | 3 | 5
Neutrophil count decreased (Investigations) | 10 | 7 | 1 | 0
Platelet count decreased (Investigations) | 19 | 9 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 0 | 2
Weight loss (Investigations) | 10 | 13 | 2 | 4
White blood cell decreased (Investigations) | 15 | 9 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 18 | 22 | 5 | 7
Dehydration (Metabolism and nutrition disorders) | 7 | 3 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 11 | 6 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 7 | 4 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 11 | 6 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 14 | 5 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 7 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 8 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 7 | 6 | 1 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 14 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8 | 2 | 3
Dizziness (Nervous system disorders) | 7 | 3 | 2 | 5
Dysgeusia (Nervous system disorders) | 15 | 19 | 9 | 2
Headache (Nervous system disorders) | 7 | 11 | 1 | 4
Nervous system disorders-Other (Nervous system disorders) | 1 | 3 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 7 | 3 | 1
Tremor (Nervous system disorders) | 1 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 5 | 4 | 1 | 0
Depression (Psychiatric disorders) | 6 | 4 | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 5 | 0 | 1
Hematuria (Renal and urinary disorders) | 10 | 8 | 0 | 1
Proteinuria (Renal and urinary disorders) | 7 | 10 | 0 | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 2 | 5 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 4 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 13 | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 21 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 5 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 9 | 2 | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9 | 5 | 2 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 21 | 29 | 4 | 9
Hypotension (Vascular disorders) | 1 | 3 | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02761057/Prot_SAP_000.pdf